CLINICAL TRIAL: NCT06114394
Title: Analysis of the Complications in Palatal Graft Harvesting With the UPV/EHU Technique vs. Single Incision Technique.
Brief Title: Complications Related to Palatal Graft Harvesting
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Principal Investigator, Ana María García de la Fuente, Professor, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023_01
Record Dates: First submitted 2023-10-28; First posted 2023-11-02 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Cicatrization
Keywords: pain; connective tissue; palate
MeSH Terms: conditions — Cicatrix; Pain

STUDY DESIGN:
Intervention Model Description: We will perform the experimental or control technique according to the randomization sequence.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant: Initially, the subject will not know what technique has been received, the complete information regarding the surgical technique used, as the results obtained in his case, will be given in the last visit of the year.
  Observer: Another periodoncist (R.E.), outside the intervention, would be in charge of recording the clinical parameters.
  Analyst: The statistician (X.M.) does not know which treatment corresponds to each variable.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UPV/EHU technique (Aguirre-Zorzano et al 2017) (Experimental): Harvesting a connective tissue graft from palate by the UPV/EHU technique.
  Interventions: Procedure: UPV/EHU technique (Aguirre-Zorzano et al 2017)
- Single incision technique (Huerzeler & Weng 1999) (Active Comparator): Harvesting a connective tissue graft from palate by the single incision technique
  Interventions: Procedure: Single incision technique (Huerzeler & Weng 1999)

INTERVENTIONS:
Procedure: UPV/EHU technique (Aguirre-Zorzano et al 2017) — The "UPV/EHU technique" (Aguirre-Zorzano et al., 2017) begins with the elevation of the full thickness flap (FTF) in the palate and an intrasulcular incision performed with a number 12 blade, preserving the papillae in the interproximal spaces. Then, the FTF is dissected with a 15c blade, holding the flap with tissue forceps, leaving the epithelium and a thin layer of the connective tissue in the flap, so that the underlying connective tissue can be harvested. After that the flap is sutured.
  Arms: UPV/EHU technique (Aguirre-Zorzano et al 2017)
Procedure: Single incision technique (Huerzeler & Weng 1999) — The CTG is harvested with the single incsion technique described by Huerzeler & Weng in 1999.
  Arms: Single incision technique (Huerzeler & Weng 1999)

SUMMARY:
Soft tissue defects can be a problem, especially in patients with high smile lines; in these clinical scenarios, the treatment with periodontal plastic surgery in combination with the use of a connective tissue graft (CTG) is considered the gold-standard procedure.

Single incision technique (Huerzeler & Weng, 1999) is one of the suggested procedures to harvest the CTG from palate. The UPV/EHU technique (Aguirre-Zorzano et al, 2017) showed less inflammation and post-surgical complications than trap-door technique, but also other technique should to be analysed.

However, there is still no consensus about which is the best technique to obtain this kind of graft. Therefore, clinicians should justify their choice based on the tissue's quality obtained and the patient's well-being, producing the least number of complications, such as inflammation, post-surgical pain, or recession in the donor area.

HYPOTHESIS:

Does the technique of obtaining an CTG of the palate using the "UPV/EHU technique" (Aguirre-Zorzano et al., 2017) result in a lower number of complications versus the "single incision technique" (Huerzeler & Weng, 1999)?

OBJECTIVES The main objective is to assess whether the complications occurring with the harvesting of the CTG using the "UPV/EHU technique" (Aguirre-Zorzano et al., 2017) are lower than with the "single incision technique"(Huerzeler & Weng, 1999), knowing the patient's perception of pain.

The secondary objectives are: a) necrosis of the palate, b) possible resulting recession in the donor area, and c) characteristics of the graft obtained

DETAILED DESCRIPTION:
Type of Study: randomized clinical trial

Two different treatments (UPV/EHU technique (test) (Aguirre-Zorzano et al. 2017) vs. Single Incision technique (control) (Huerzeler & Weng, 1999)) will be compared. These techniques are usually used to harvest a CTG from the palate.

Main outcome: complications in the donor area.

Follow-up: 6 months.

UNIT OF ANALYSIS: The patient of the Master's Degree in Periodontology and Osseointegration from the University of the Basque Country (UPV/EHU), requires treatment with a CTG harvested from the palate.

SAMPLE SIZE CALCULATION: Using the visual analog pain scale (VAS pain) as the primary response variable, it is estimated that, to find a difference of 1 between test and control, with an SD= 1.26 (Wessel & Tatakis 2008), an alpha risk of 5% and a power of 85%, we would need 29 patients for each treatment group (Domenech and Granero 2010). In addition, taking into account possible dropouts, we would increase the number of patients by 20%, finally recruiting 35 patients per group.

Statistical analysis:

A descriptive study of the sample will be performed, based on moments (mean, standard deviation) if the parameters of normality are met or on ordinations (median and interquartile range), in case the parameters of normality are not met.

Subsequently, analytical statistics will be performed, and in addition, the intensity and duration of post-surgical pain after each surgical technique adjusted for possible confounding factors (clinical level of central sensitization, presence of pre-surgical pain, presence of post-surgical complications, use of added analgesic treatment) will be assessed using logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the UPV/EHU university dental clinic who required a connective graft of the palate in their treatment.
* Patients ≥ 18 years-old
* Absence of active periodontal disease ( healthy periodontal patients or periodontal patients who had received active periodontal treatment, and now they are included in a tailored supportive periodontal program)
* Full-mouth plaque index (FMPI) (O'Leary y cols. 1972) and full-mouth bleeding index (FMBI) (Ainamo y Bay, 1975) ≤ 25%

Exclusion Criteria:

* Smokers of ≥ 10 cigarettes/day
* Systemic conditions that contraindicated surgery
* The use of analgesic and/or anti-inflammatory drugs in the last 72 h
* The use of opioid drugs, anticonvulsants and/or antidepressants, except selective serotonin inhibitors, i.e., those drugs that act by reducing the painful experience
* Pregnancy or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-12-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Post-surgical pain perception | After surgery up to 14 days
  The subject will we instructed to collect their perception of post-surgical pain in the VAS based on the UPV/EHU Pain diary (Fernandez-Jimenez et al, 2021). Specifically the subject will record: Its intensity (0-100mm), its duration (minutes or hours) and if any analgesic treatment has been necessary (No o Yes: Which?).

SECONDARY OUTCOMES:
Central Sensitization Inventory severity-level score of the subject Central Sensitization inventory (CSI) (Mayer et al. 2012) | Baseline
  Central Sensitization inventory (CSI) (Mayer et al. 2012) will be done, in which each subject will be asked on the frequency in which he perceives 25 symptoms and will be given a score of 0-4 finally establishing a clinical level in a range of 0-100 points (Subclinical: 0-29; Medium: 30-39; Moderate: 40-49 ; Severe: 50-59; Extreme: 60-100).
Pre-surgical pain perception. | Baseline
  In the VAS based on the UPV/EHU Pain Diary (Fernandez-Jimenez et al 2021) the examiner will record if the subject has had regional head and neck pain in the last month and if there is any pain in the immediate preoperative, if it is affirmative the intensity will be noted
Necrosis of the palate | up to 7 days post-srugery
  After using 2 CP-11 periodontal probes by placing them perpendicularly, thus obtaining a measured in the X-axis and another in the Y-axis and multiplying both results, the donor area in mm2 will be obtained. From that point on, it will be possible to determine what degree of necrosis has occurred in the donor area by taking the following values as a reference (Aguirre-Zorzano et al. 2017):
  Value 0: total absence of necrosis. Value 1 : ≦30% of the donor area. Value 2: ≧ 30% of the donor area.
Gingival recession (REC) in donor area | Change from baseline at following surgery sixth month respectively.
  Distance in mm from the amelocementaria line the gingival margin, measured at the vestibular midpoint. It will be registered in all the teeth present in the donor area at the beginning, and, during the follow-up only in the recessions to be treated
Post-surgical complications | After surgery first seven days.
  The presence or not, as the description, of the post-surgical complications (PSC) that may appear will be collected.
Thickness of the donor area of the palate and of the connective tissue graft | Surgery
  measured using 2 CP-11 periodontal probes and placing them perpendicularly, thus creating a measurement in the X axis and another in the Y axis, in order to obtain the area in mm2 of the graft obtained by multiplying both measurements, and placing a file with a rubber stopper in the central area of the graft to measure its thickness.
Length of the donor area of the palate and of the obtained CTG(mm) | Surgery
  by positioning a CP-11 periodontal probe parallel to the donor area on the palate, as well as on the connective tissue graft obtained
Width of the donor area of the palate and of the obtained CTG (mm) | Surgery
  by positioning a CP-11 periodontal probe perpendicular to the donor area on the palate, as well as on the obtained connective tissue graft.
Area (mm2) of the donor area of the palate and of the obtained CTG | Surgery
  : measurement obtained by multiplying the variables length and width of the donor area, as well as of the obtained CTG.
Extension of the bed recipient. | Baseline
  The number of teeth or implants will be registered in the bed receipt.
Full mouth bleeding index (FMBI) (Aynamo & Bay, 1975) | Change from baseline at following surgery sixth month respectively.
  After a periodontal probing of all teeth, the presence (yes or no) of bleeding is recorded dichotomously at 6 points per tooth (mesio-bucal, mid-bucal, disto-bucal, mesio-lingual, mid-lingual and disto-lingual) and the percentage of sites that bleed from the total of probed sites is calculated (Ainamo and Bay 1975)
Full mouth plaque index (FMPI). | Change from baseline at following surgery sixth month respectively.
  A plaque developer is used and the presence (yes or no) of plaque is recorded dichotomously at 6 points per tooth (mesio-bucal, mid-bucal, disto-bucal, mesio-lingual, mid-lingual and disto-lingual) and the percentage of sites with plaque of the total probed sites is calculated (O'Leary et al 1972).
Probing depth (PD) | Change from baseline at following surgery sixth month respectively.
  Distance in millimeters from the gingival margin to the bottom of the periodontal pocket. It will be recorded at the beginning in all teeth present (except wisdow teeth) in 6 points per tooth (mesio-bucal, mid-bucal, disto-bucal, mesio-lingual, mid-lingual and disto-lingual) and, during follow-up, only in the recessions to be treated at the vestibular mid-point.

CONTACTS AND LOCATIONS:
Overall Officials: ANA MARIA GARCIA DE LA FUENTE, PHD, Study Director — UPV/EHU
Locations (1):
- UPV/EHU, Leioa, Vizcaya, Spain

REFERENCES:
- [Background] Zucchelli G, Mounssif I, Mazzotti C, Montebugnoli L, Sangiorgi M, Mele M, Stefanini M. Does the dimension of the graft influence patient morbidity and root coverage outcomes? A randomized controlled clinical trial. J Clin Periodontol. 2014 Jul;41(7):708-16. doi: 10.1111/jcpe.12256. Epub 2014 May 8. PMID 24708394
- [Result] Del Pizzo M, Modica F, Bethaz N, Priotto P, Romagnoli R. The connective tissue graft: a comparative clinical evaluation of wound healing at the palatal donor site. A preliminary study. J Clin Periodontol. 2002 Sep;29(9):848-54. doi: 10.1034/j.1600-051x.2002.290910.x. PMID 12423299
- [Result] Harris RJ, Miller R, Miller LH, Harris C. Complications with surgical procedures utilizing connective tissue grafts: a follow-up of 500 consecutively treated cases. Int J Periodontics Restorative Dent. 2005 Oct;25(5):449-59. PMID 16250567
- [Result] Griffin TJ, Cheung WS, Zavras AI, Damoulis PD. Postoperative complications following gingival augmentation procedures. J Periodontol. 2006 Dec;77(12):2070-9. doi: 10.1902/jop.2006.050296. PMID 17209793
- [Result] Hurzeler MB, Weng D. A single-incision technique to harvest subepithelial connective tissue grafts from the palate. Int J Periodontics Restorative Dent. 1999 Jun;19(3):279-87. PMID 10635174
- [Result] Aguirre-Zorzano LA, Garcia-De La Fuente AM, Estefania-Fresco R, Marichalar-Mendia X. Complications of harvesting a connective tissue graft from the palate. A retrospective study and description of a new technique. J Clin Exp Dent. 2017 Dec 1;9(12):e1439-e1445. doi: 10.4317/jced.54337. eCollection 2017 Dec. PMID 29410760
- [Result] Zucchelli G, Mele M, Stefanini M, Mazzotti C, Marzadori M, Montebugnoli L, de Sanctis M. Patient morbidity and root coverage outcome after subepithelial connective tissue and de-epithelialized grafts: a comparative randomized-controlled clinical trial. J Clin Periodontol. 2010 Aug 1;37(8):728-38. doi: 10.1111/j.1600-051X.2010.01550.x. Epub 2010 Jun 24. PMID 20590963